CLINICAL TRIAL: NCT04136210
Title: Perioperative Clinical, Hemodynamic Data and Prognosis Assessment in Patients Who Undergo Cardiovascular Surgery; Registry Construction
Brief Title: Registry Construction for Perioperative Data in Patients Undergoing Cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Other Study IDs: Heart Registry
Record Dates: First submitted 2019-10-13; First posted 2019-10-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this registry is to obtain perioperative data in patients undergoing cardiac or thoracic aortic surgery and find out relations between the data and investigate several causes affecting postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac or thoracic aortic surgery

Exclusion Criteria:

* refused to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac or thoracic aortic surgery
Sampling Method: Non-Probability Sample
Enrollment: 1568 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics | Before surgery
  1. Sex
  2. Age
  3. Height
  4. Weight
  5. Body mass index
  6. Underlying disease Family history
  7. Previous operation history
  8. Current medication Preoperative hemodialysis
  9. Preoperative cardiopulmonary resuscitation
  10. Preoperative mechanical ventilation
  11. Preoperative intra-aortic balloon pump
  12. Preoperative intravenous drug and dose
  13. Alcohol history, smoking history
  14. Drug allergy
  15. Functional capacity, ASA classification, NYHA class
  16. EuroSCORE, STS score, SOFA score
Preoperative data | Before surgery
  1. Vital sign including systolic blood pressure, diastolic blood pressure, mean blood pressure, pulse pressure, heart rate, SpO2, body temperature, consciousness, GCS (Glasgow Coma Scale), central venous pressure, pulmonary arterial pressure, and respiratory rate
  2. Laboratory data including CBC (Hb, Hct, WBC, platelet), Electrolyte (Na, K, Ca, Mg), coagulation (PT INR, aPTT, fibrinogen), ABGA (Hct, pH, pCO2, pO2, HCO3-, BE, SaO2), BUN/Creatinine, OT/PT, Total bilirubin, CRP, cardiac enzyme (Troponin I, CK, CK-MB), albumin, glucose, HbA1C, lactate, and creatinine clearance
  3. ABGA (Hct, pH, pCO2, pO2, HCO3-, BE, SaO2, Na, K, iCa, Glucose, Lactic acid)
  4. Imaging data including chest X-ray, chest CT, Brain MRI/A, coronary angiography, CT angiography, cardiac MRI, myocardiac SPECT, and abdomen CT
  5. ECG (rhythm, QTc interval), PFT, Echocardiography (Ejection fraction, RWMA, Pulmonary HTN, Valve abnormality), and esophagogastroduodenoscopy
Intraoperative and postoperative data | During surgery and until 48 hours after surgery
  1. Vital sign
  2. ECG analysis
  3. Stroke volume variation, pulse pressure variation
  4. Cardiac index, cardiac output, stroke volume, mixed venous oxygen saturation
  5. Airway and respiratory indicators
  6. Bispectral index
  7. Patient state index (PSi)
  8. Tissue oxygen saturation of brain and limbs
  9. Tissue oxygen saturation (StO2) during vascular occlusion test (VOT)
  10. Transcutaneous CO2 (PtcCO2), transcutaneous O2 (PtcO2)
  11. Sublingual SDF imaging (MicroScan; MicroVision Medical, Amsterdam, the Netherlands)
  12. Pupil reactivity assessment scale
  13. Coagulation: ROTEM, Multiplate
  14. Laboratory data
  15. ABGA
  16. Cardiac enzyme
Operation data | During surgery
  1. Type of operation
  2. Emergency or elective
  3. Types and doses of anesthetics, anesthesia time, surgery time
  4. Location of arterial lines
  5. Infused fluid and dose, estimated blood loss, blood transfusion, and urine output
  6. Coronary artery bypass surgery: type of bypass artery, bypass time for each artery
  7. Cardiopulmonary bypass A. Cardiopulmonary bypass protocol B. Types and doses of used drug, rewarming time, duration of CPB, time of aortic clamping, transfusion dose
  8. Aortic arch surgery: total circulatory arrest, circulatory arrest duration, cerebral perfusion
  9. Intraoperative TEE finding
  10. Assist device including IABP, ECMO, LVAD, and RVAD
  11. Rescue drug usage and dose
  12. Tranexamic acid and vitamin K usage
  13. Drug reaction or specific event
Postoperative ICU data | 1 year after surgery
  1. Imaging data including chest X-ray, chest CT, Brain MR/CT, Echocardiography
  2. Mechanical ventilation duration
  3. ICU stay duration
  4. Hospital stay duration
  5. Postoperative pain control, sedatives
  6. Drug usage and dose (Epinephrine, norepinephrine, dobutamine, dopamine, milrinone, vasopressin, nitroglycerin, phenylephrine, calcium chloride, lidocaine, amiodarone, digoxin, diltiazem, bicarbonate, and adenosine)
  7. Assist device including IABP, ECMO, LVAD, and RVAD
  8. Infused fluid and dose (crystalloid, colloid), estimated blood loss, blood transfusion (RBC, FFP, Platelet, cryoprecipitate, self-blood salvage), urine output at ICU admission, 24 hours / 48 hours after ICU admission.
Complications | 1 year after surgery
  1. Cardiac complications
  2. Respiratory complications
  3. Neurologic complications
  4. Renal complications
  5. Infectious complications
  6. Gastrointestinal complications
  7. Adverse drug reaction
  8. Bleeding complications
  9. Thrombotic complications
  10. Postoperative multiorgan failure (SOFA score)
  11. Mortality including in hospital mortality
  12. Re-operation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Jung DE, Park D, Kim TJ, Lee HC, Bae J, Nam K, Jeon Y, Cho YJ. Intraoperative neurological pupil index and postoperative delirium and neurologic adverse events after cardiac surgery: an observational study. Sci Rep. 2023 Aug 24;13(1):13838. doi: 10.1038/s41598-023-41151-z. PMID 37620412